CLINICAL TRIAL: NCT04790240
Title: The Trial Uses Medicinal Herbs to Direct T Cells to Engulf the COVID-19 Virus and Protect the Organs Well
Brief Title: Medical Herbs Inhibit Inflammation Directing T Cells to Kill the COVID-19 Virus (COVID)
Acronym: COVID
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: All Natural Medicine Clinic, LLC (Other)
Responsible Party: Principal Investigator, Wanzhu Hou, President, All Natural Medicine Clinic, LLC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHM2282395-1
Record Dates: First submitted 2021-02-23; First posted 2021-03-10 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Covid19 Virus Infection
Keywords: Medicinal Herbs; Virus; COVID-19; Coronavirus Disease 2019; Infections; Inflammation; Immunity; Metabolite; clots; thrombus; Viral Pneumonia; Fever; Cough; Chest congestion
MeSH Terms: conditions — COVID-19; Virus Diseases; Infections; Inflammation; Thrombosis; Pneumonia, Viral; Fever; Cough | interventions — Standard of Care; Dosage Forms

STUDY DESIGN:
Intervention Model Description: The participants are randomly divided into two groups: the treatment group and the control group. Both groups receive the same medications, but the treatment group also receives medical herbs to compare both groups' differences on their symptoms and blood data, virus marks.
Who Masked: Participant, Care Provider
Masking Description: The participants will be randomly divided into two groups by computer. The conventional practitioners who prescribe medications for the participants will not know who will go to the treatment group. Participants will know which group they are in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Inflammation (I) (Active Comparator): 1. Upper respiratory inflammation.
  2. Fever.
  3. Lower respiration inflammation.
  Interventions: Dietary Supplement: Inflammation (I); Drug: Standard of care
- Inflammation (II) (Active Comparator): Cough, chest pain
  Interventions: Dietary Supplement: Inflammation (II); Drug: Standard of care
- Inflammation (III) (Active Comparator): 1. Metabolites
  2. Clots
  Interventions: Dietary Supplement: Inflammation (III); Drug: Standard of care

INTERVENTIONS:
Dietary Supplement: Inflammation (I) — 1. upper respiratory inflammation (PurInf (I)): Lonicerae Flos 2.4g, Forsythiae Fructus 2.4g, Schizonepetae Herba 2g, Saposhnikoviae Radix 2g, Cicadae Periostracum 1g, Sophorae flavescentis Radix 2.4g, Atractylodis Rhizoma 2g, Angelicae dahuricae Radix 2g, Menthae haplocalycis Herba 2g, Arctii Fructus 2g, Glycyrrhizae Radix 1g
  2. high fever (PurInf (II)): Bupleuri Radix 3g, Scutellariae Radix 2.4g, Gypsum fibrosum 4g, Anemarrhenae Rhizoma 3g
  3. lower Respiratory system inflammation (PurInf (III)): Scutellariae Radix 2.4g, Coptidis Rhizoma 1g, Phellodendri Cortex 2.4g, Gardeniae Fructus 2.4g, Houttuyniae Herba 4g, Golden Buckwheat 3g
  Other Names: PurInf (I), PurInf (II), PurInf(III)
  Arms: Inflammation (I)
Dietary Supplement: Inflammation (II) — Platycodi Radix 2.4g, Peucedani Radix 2.4g, Cynanchi stauntonii Rhizoma 2.4g, Asteris Radix 2.4g, Stemonae Radix 2.4g, Lepidii Descurainiae Semen 2.4g, Plantaginis Semen 2.4g
  Other Names: PurCo
  Arms: Inflammation (II)
Dietary Supplement: Inflammation (III) — 1. Metabolites, abnormal fluids (PurPhl):
     Citri reticulatae Pericarpium 1.2g, Citri grandis Exocartium rubrum 2g, Aurantii Fructus immaturu 2g, Pinelliae Rhizoma preparatum 2.4g, Arisaematis Rhizoma preparatum 2.4g, Amoni Fructus 1g, Trichosanthis Fructus 2.4g, Fritillatiae cirrhosae Bulbu 2.4g, Poria 2.4g, Rhei Radix et Rhizoma 1g
  2. Capillaries circulation disorder (PurClo):
  Salviae miltiorrhizae Radix 2.4g, Curcumae Radix 2.4g, Paeoniae Radix rubra 2.4g, Persicae Semen 2.4g, Carthami Flos 2.4g
  Other Names: PurPhl, PurClo
  Arms: Inflammation (III)
Drug: Standard of care — remdesivir (Veklury), Colchicine, anti-SARS-CoV-2 monoclonal antibodies, bamlanivimab, Casirivimab & Imdevimab.
  Other Names: Medications

SUMMARY:
The human immune system is designed to protect individuals from external sources of infection and internal cell mutation. It works effectively and efficiently until inflammation disturbs its functioning. Once compromised by inflammation, the immune system loses its capacity to recognize antigens and dependably defend the body against disease and illness.

When COVID-19 invades humans, it causes an immune-storm (cytokine-storm) that can directly damage the organ(s), leading to death. The virus is an antigen - a trigger - but it is not the actual reason that causes organ failure and death; instead, it is the body's over immune reaction that is the cause. In attempting to protect the body, the immune system overreacts to the antigen, which includes the infected cells, which causes a cytokine-storm, and the subsequent and rapid shut down of the infected individual's organ(s)' structure, leaving the body without sufficient strength or time to fight back. When the medical herbs join the body, it can slow down the immune reaction. Medical herbs benefit the physical body; they protect the cells and organism structure and mediate the immune response, allowing the T cells to kill the virus (mutated or not) internally. Such success has been achieved by the All Natural Medicine Clinic during pre-clinical trials.

This clinical study's goal is to demonstrate that the immune system can be rebuilt and retrained, using natural medicine (i.e., medical herbs), to kill the virus without causing the immune storm, and to explore the mechanism by which these medical herbs, which have been used for thousands of years for healing, achieve results.

DETAILED DESCRIPTION:
According to CDC data, as of January 30, 2021, 25,780,144 individuals residing in the United States had been infected by COVID-19 and 435,151 had died as a result of the disease. No drug has yet been identified that explicitly kills the COVID-19 virus. While various vaccines have been developed to prevent infection, the virus continues to mutate, and scientific research remains behind the virus trajectory.

The human immune system, when functioning properly, can prevent the body from succumbing to infections from external sources and from internal cell mutations, including the COVID-19 virus and cancer cells. That is, the defense system comes from nature. This clinical study proves that the immune system can respond to those antigens and kill them if the immune system is given a chance. However, the human immune system can become compromised through inflammation and subsequently unable to successfully prevent infection and cancer.

When COVID-19 invades humans, it causes an immune-storm (cytokine-storm) that can directly damage the organ(s), leading to death. The virus is an antigen - a trigger - but it is not the actual reason that causes organ failure and death; instead, it is the body's over-immune reaction that is the cause. In attempting to protect the body, the immune system overreacts to the antigen, which includes the infected cells, which causes a cytokine-storm, and the subsequent and rapid shut down of the infected individual's organ(s)' structure, leaving the body without sufficient strength or time to fight back.

Medical herbs can mediate the immunity disorder caused by infections, and mutated cells, including COVID-19 and its mutations. Our pre-clinical study found that the medical herbs inhibit the inflammation expression, reduce the chance of cytokine-storm, prevent deterioration, and reduce the mortality rate. In addition, the T cells can perform their job when the inflammation is under control. The virus and cancer cells belong to antigens that should be killed by natural killer (NK) cells and T cells. This clinical study aims not to provide drugs to kill the antigens, but rather to create the necessary conditions inside the human body to allow the immune system a chance to overcome the antigens. The clinic has used this treatment concept to successfully treat infected patients and cancer patients.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study if any of the following criteria apply:

* Individuals diagnosed with COVID-19 virus infection in the past 1-20 days must submit the proved metrics of COVID-19 virus marks positive during the registration;
* The age of participants is between 10-70 years old;
* The participants are received or not received conventional medication treatment, and continuing the treatment patients, could be enrolled in this clinical study;
* This clinical study is not restricted to gender, age, sex, race, and nationality;
* The participants must have reports of CBC, C3, C4, IgM, IgG, CD4/CD8, and lungs' images ready before the clinical study;
* The Participants must repeat the evaluation experiment during and at the end of the clinical study.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Individuals with a prior COVID-19 virus infection that no longer shows up from COVID-19 testing;
* Children who are younger than 10-year-old, cannot control themselves to take the medical herbs on time;
* Elders whose age beyond 70-year-old, with severe underline illness;
* COVID-19 virus-infected patients who do not feel willing to take medical herbs;
* Patients diagnosed with COVID-19 virus infection cannot consistently finish the treatment courses for a specific reason;
* Patients diagnosed with COVID-19 virus infection but do not willing to share their information with the public;
* Current or past participation within a specified timeframe in another clinical trial, as warranted by this intervention's administration;
* Severe patients, when there have insufficient normal cells, can be adjusted, with pre-list diseases life-threatening.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
recovering damaged organ | 3 weeks
  comparing imagen of lungs
inhibiting inflammation | 3 weeks
  comparing C-reactive protein (CRP)
preventing the antibody depositing on antigen | 6 weeks
  measuring complement: C3, C4

SECONDARY OUTCOMES:
monitoring the antibody level | 6 weeks
  measuring immunoglobulin M (IgM), immunoglobulin G (IgG)
correcting reversed immunity ratio | 6 weeks
  measuring cluster of differentiation 4/cluster of differentiation 8 (CD4/CD8)
tracking the COVID virus marks | 3 weeks
  SARS-CoV-2 Diagnostic (Molecular or Antigen) Testing

CONTACTS AND LOCATIONS:
Overall Officials: Wanzhu Hou, CMD,MD(CN), Principal Investigator — All Natural Medicine Clinic, LLC
Locations (1):
- All Natural Medicine Clinic, LLC, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
When we finish the project of the clinical study, we will share the individual participant's data (IPD) (but is not personal private to share) when the results in the publication
Supporting Information: Study Protocol
Time Frame: The clinical study may start on February 1, 2021; the ending of the say maybe is December 31, 2022. The IPD sharing will begin after the publication in six months.
Access Criteria: Viruses, including COVID-19, are highly likely to mutate. This capacity makes it particularly challenging to kill the virus with drugs. This clinical study designed two groups, both of they used the same drugs, but the treatment group pluses medical herbs, then both groups parallelly receive the treatment, then compare participants symptoms, blood test of immunity, the lungs imagine, and COVID-19 virus index, the difference in both group, analysis the symptoms and the mechanism.
URL: http://www.anmedicine.com

REFERENCES:
- [Background] Wannzhu Hou Cellular Structure and its Function is the key for heeling Diseases, Certification and Registration number: TXu 1-938-144 July 30, 2014
- [Background] Rosendahl Huber S, van Beek J, de Jonge J, Luytjes W, van Baarle D. T cell responses to viral infections - opportunities for Peptide vaccination. Front Immunol. 2014 Apr 16;5:171. doi: 10.3389/fimmu.2014.00171. eCollection 2014. PMID 24795718
- [Background] Zhou LK, Zhou Z, Jiang XM, Zheng Y, Chen X, Fu Z, Xiao G, Zhang CY, Zhang LK, Yi Y. Absorbed plant MIR2911 in honeysuckle decoction inhibits SARS-CoV-2 replication and accelerates the negative conversion of infected patients. Cell Discov. 2020 Aug 5;6(1):54. doi: 10.1038/s41421-020-00197-3. eCollection 2020. No abstract available. PMID 32802404
- [Background] Peters M. Actions of cytokines on the immune response and viral interactions: an overview. Hepatology. 1996 Apr;23(4):909-16. doi: 10.1053/jhep.1996.v23.ajhep0230909. No abstract available. PMID 8666349
- [Background] Zhou H, Sun L, Yang XL, Schimmel P. ATP-directed capture of bioactive herbal-based medicine on human tRNA synthetase. Nature. 2013 Feb 7;494(7435):121-4. doi: 10.1038/nature11774. Epub 2012 Dec 23. PMID 23263184
- [Background] Dosch M, Gerber J, Jebbawi F, Beldi G. Mechanisms of ATP Release by Inflammatory Cells. Int J Mol Sci. 2018 Apr 18;19(4):1222. doi: 10.3390/ijms19041222. PMID 29669994
- [Background] Chen RJ, Jinn TR, Chen YC, Chung TY, Yang WH, Tzen JT. Active ingredients in Chinese medicines promoting blood circulation as Na+/K+ -ATPase inhibitors. Acta Pharmacol Sin. 2011 Feb;32(2):141-51. doi: 10.1038/aps.2010.197. PMID 21293466
- [Background] Samuels N. Herbal remedies and anticoagulant therapy. Thromb Haemost. 2005 Jan;93(1):3-7. doi: 10.1160/TH04-05-0285. PMID 15630483
- [Background] Soni S, O'Dea KP, Tan YY, Cho K, Abe E, Romano R, Cui J, Ma D, Sarathchandra P, Wilson MR, Takata M. ATP redirects cytokine trafficking and promotes novel membrane TNF signaling via microvesicles. FASEB J. 2019 May;33(5):6442-6455. doi: 10.1096/fj.201802386R. Epub 2019 Feb 18. PMID 30776316
- [Result] Wanzhu Hou, et al. Treating Autoimmune disease with Chinses Medicine, Elsevier, 2011
- See also: We widely treat and research infected and non-infected diseases based on recovering the damaged structure and function of cells. — http://www.anmedicine.com